CLINICAL TRIAL: NCT01284075
Title: The Effect of Guided Imagery and Music Therapy on Post-Operative Recovery After Gynecological Oncology Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low accrual
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2009NTLS051; 0912M75053 (Other: IRB, University of Minnesota)
Record Dates: First submitted 2011-01-25; First posted 2011-01-26 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2014-08

CONDITIONS: Ovarian Cancer; Uterine Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Uterine Neoplasms | interventions — Imagery, Psychotherapy; Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Guided Imagery and Music therapy group (GIMT) (Experimental): Participants will undergo a standardized regimen of peri-operative guided imagery and music therapy guided by CDs (compact disc). The peri-operative regimen will include: listening to the CD while in the pre-operative holding area, listening to the CD during the procedure; listening to the CD after the procedure beginning on the evening of post-operative day (POD)#0 and continuing twice a day until POD#3.
  Interventions: Behavioral: Guided imagery and music therapy
- White Noise Group (WN) (Active Comparator): Control group (WN) will listen to a CD with white noise. Participants' regimen will include: listening to the CD while in the pre-operative holding area, listening to the CD during the procedure; listening to the CD after the procedure beginning on the evening of post-operative day (POD)#0 and continuing twice a day until POD#3.
  Interventions: Behavioral: White Noise
- No Interventions Group (CP) (Active Comparator): Control group (CP) will have no intervention at all and will follow our current peri-operative procedures.
  Interventions: Other: No intervention

INTERVENTIONS:
Behavioral: Guided imagery and music therapy — Participants will undergo a standardized regimen of peri-operative guided imagery and music therapy guided by CDs (compact disc). The peri-operative regimen will include: listening to the CD while in the pre-operative holding area, listening to the CD during the procedure; listening to the CD after the procedure beginning on the evening of post-operative day (POD)#0 and continuing twice a day until POD#3.
  Arms: Guided Imagery and Music therapy group (GIMT)
Behavioral: White Noise — Control group (WN) will listen to a CD with white noise. Participants' regimen will include: listening to the CD while in the pre-operative holding area, listening to the CD during the procedure; listening to the CD after the procedure beginning on the evening of post-operative day (POD)#0 and continuing twice a day until POD#3.
  Arms: White Noise Group (WN)
Other: No intervention — Control group (CP) will have no intervention at all and will follow our current peri-operative procedures.
  Arms: No Interventions Group (CP)

SUMMARY:
This pilot study will be a prospective, randomized trial which will take place at the University of Minnesota Medical Center (UMMC). Eligible patients will be identified at the time of their first clinic visit. If selected to be involved in the study, the patients will be randomized to one of three different groups: a Guided Imagery and Music therapy group (GIMT) or one of two control groups.

DETAILED DESCRIPTION:
The GIMT group will undergo a standardized regimen of peri-operative guided imagery and music therapy guided by CDs. As there are no studies which discuss whether the act of listening to any therapy will affect outcomes, we will also explore whether white noise can affect outcomes as well. Therefore, one control group (WN) will abide by the same regimen and will listen to a CD with white noise; the other control group (CP) will have no intervention at all and will follow our current peri-operative procedures.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will include women who are being seen at the Women's Health Center by the Gynecological Oncology group at the University of Minnesota (UMMC). These women will be considered for inclusion based on their projected surgery: exploratory laparotomy. Subjects will have to have their surgery at the UMMC within 1 month of their clinic visit. Patients may be undergoing surgery for either known cancer (ovarian or uterine) or high suspicion for malignancy.

Exclusion Criteria:

* < 19 years old
* pregnant
* undergoing a procedure other than laparotomy
* scheduled to be discharged the same day of surgery
* chronic narcotic pain medication users
* if they are currently using or planning on using other complementary alternative medicine (CAM) therapies prior to or after surgery.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-04; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Change in Mean Pain Score | From Admission through 4 Weeks Post Surgery
  Determined by using a Visual Analog Pain Scale (VAS)- A Visual Analogue Scale (VAS) for pain is a horizontal line 100 mm in length with the left end labeled 'No pain' and the right end labeled 'Very severe pain'. The subject marks a point on the line that represents their perception of their current state. The VAS score is determined by measuring the distance from the left end of the line to the point on the line marked by the subject. The range of possible values for this pain score is 0 to 100 millimetres.

SECONDARY OUTCOMES:
Use of Pain Medication | From Admission to 4 Weeks Post Surgery
  List of pain medications and number of times administered.
Use of Anti-Nausea Medications | From Admission to 4 Weeks Post Surgery
  List of anti-emetic medications and number of times administered
Mean Change in Patient Quality of Life Score | From Admission to 4 Weeks Post Surgery
  Using the Functional Assessment of Cancer Therapy General Scale (FACT-G) for patients with cancer (consisting of a four-factor structure - "Physical well-being", "Social-family well-being", "Functional well-being" and "Emotional well-being"). Five response choices range from "not at all" to "very much".
Average Number of Days Hospitalized | From Admission through 4 Weeks Post Surgery
Hospital Readmission Rates | From Admission Through 4 Weeks Post Surgery
Change in Profile of Mood States (POMS) | From Admission Through 4 Weeks Post Surgery
  The Profile of Mood States (POMS) original scale contains 65 self-report items using the 5-point Likert Scale. Participants can choose from 0 (not at all) to 4 (extremely). The test takes approximately 3 to 7 minutes for healthy participants, and longer for the physically ill.
Length of Hospital Stay (Days) | From Admission through 4 Weeks Post Surgery

CONTACTS AND LOCATIONS:
Overall Officials: Amy Jonson, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States